CLINICAL TRIAL: NCT00721773
Title: Effects of Benazepril,Valsartan or Combination of Both on Residual Renal Function in Peritoneal Dialysis Patients
Brief Title: Renal Protective Effects of Renin Angiotensin System (RAS) Inhibitor in Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xue Qing Yu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDRRF
Record Dates: First submitted 2008-07-22; First posted 2008-07-24 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Renal Function Disorder
Keywords: Continuous Ambulatory Peritoneal Dialysis; Angiotensin-converting Enzyme Inhibitor; Angiotensin II Receptor Blocker; Renin angiotensin system inhibitor; Residual Renal Function
MeSH Terms: interventions — benazepril; Valsartan; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ACE inhibitor, benazepril (Experimental): Benazepril will be started at 10 mg/day and will be up-titrated to 20 mg/day according to BP control and tolerability.
  Interventions: Drug: Benazepril
- Angiotensin receptor blocker, valsartan (Experimental): Valsartan will be started at 80 mg/day and will be up-titrated to 160 mg/day according to BP control and tolerability.
  Interventions: Drug: Valsartan
- RAS inhibitors, benazepril+valsartan (Experimental): Benazepril will be started at 10 mg/day and will be up-titrated to 20 mg/day, and valsartan will be started at 80 mg/day and will be up-titrated to 160 mg/day according to BP control and tolerability.
  Interventions: Drug: Benazepril+Valsartan
- non-RAS inhibitors, control (Active Comparator): Drug: antihypertensive agents, except ACE inhibitors and ARBs. Administration of antihypertensive agents will select as follows: CCB→β-blocker→α-blocker.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Benazepril — Patients with hypertension will take 10-20mg benazepril per day, antihypertensive agents other than ACE inhibitors and ARBs will be allowed. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 120-140/70-90 mmHg.
  Other Names: Benazepril group
  Arms: ACE inhibitor, benazepril
Drug: Valsartan — Patients with hypertension will take 80-160mg valsartan per day, antihypertensive agents other than ACE inhibitors and ARBs will be allowed. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 120-140/70-90 mmHg.
  Other Names: Valsartan group
  Arms: Angiotensin receptor blocker, valsartan
Drug: Benazepril+Valsartan — Patients with hypertension will take 10-20mg benazepril plus 80-160mg valsartan per day, antihypertensive agents other than ACE inhibitors and ARBs will be allowed. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 120-140/70-90 mmHg.
  Other Names: Benazepril plus Valsartan group
  Arms: RAS inhibitors, benazepril+valsartan
Drug: Control — Patients in the control group will administer antihypertensive agents, except ACE inhibitors and ARBs. Doses are adjusted appropriately to achieve and maintain the target blood pressure of 120-140/70-90 mmHg.
  Other Names: Control group
  Arms: non-RAS inhibitors, control

SUMMARY:
This is a multicentre study examining the effectiveness of angiotension converting enzyme inhibitor (ACEI), angiotensin receptor blocker (ARB) or a combination of both in reducing the rate of decline in residual renal function (RRF) in continuous ambulatory peritoneal dialysis (CAPD) patients.

DETAILED DESCRIPTION:
RRF has been shown to decline progressively with time on dialysis in both CAPD and hemodialysis. Although RRF is an important determinant of mortality and morbidity in peritoneal dialysis (PD) patients, few studies have addressed therapeutic approaches for preserving RRF after the initiation of dialysis therapy. Blockade of the renin-angiotensin system by ACEI or ARB is a well-established approach for renoprotection in pre-dialysis chronic kidney disease patients. Up to now, only two trials showed that an ACEI, ramipril, and ARB, valsartan , were effective in the preservation of RRF of CAPD patients. However it is important to point out that the evidence cited has limitations. First, the trial only involved patients from one university teaching hospital. Second, transport characteristics, were not assessed before the start of the study. Third, the trial was too small to detect potentially important differences in health care use and survival between groups. Therefore, whether both ACEI and ARB preserve RRF, improve clinical outcomes and decrease health care use and costs should be tested in much longer and larger studies involving multiple sites. In order to confirm these findings, here the investigators will perform prospective, randomized, open-label and multiple center study to address long-term effects of ACEI, ARB and combination of both therapy on RRF in Patients on CAPD.

ELIGIBILITY:
Inclusion Criteria:

* All patients received CAPD more than 1 months
* Subjects of either sex, 20-75 years old
* Residual GFR of 3mL/min per 1.73 m2 or more
* With hypertension
* No history of taking an ACE inhibitor or angiotensin-receptor blockers for at least 1 month
* Provision of written informed consent by subject or guardian

Exclusion Criteria:

* Underlying medical conditions, such as congestive heart failure, or therapy with an ACE inhibitor or ARB
* Peritonitis or volume overload within the preceding 1 month
* Myocardial infarction within the preceding 6 months
* Clinically significant valvular disease
* Malignant hypertension
* History of hypertensive encephalopathy or cerebrovascular accident within the preceding 6 months
* Any condition that may have precluded a patient from remaining in the study, such as alcohol or drug abuse, chronic liver disease, malignant disease, or psychiatric disorder
* History of allergy or intolerance to an ACE inhibitor or ARB
* Participation in another clinic trial within 2 weeks prior to screening

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The longitudinal change in residual glomerular filtration rate (GFR) | 3 years
  Residual GFR is defined as the average of 24-hour urinary urea and creatinine clearances.

SECONDARY OUTCOMES:
Dialysis adequacy | 3 years
  Indices of the adequacy of dialysis include Kt/V and weekly creatinine clearance assessed by 24-hour dialysate and urinary collection.
Peritoneal membrane function | 3 years
  Peritoneal membrane function assessed by standard peritoneal equilibration test.
Blood pressure | 3 years
  Office systolic and diastolic blood pressure measurement during follow up period.
The time to anuria | 3 years
  Anuria is defined as urine volume < 100ml/d.
Number of participants not alive | 3 years
  Death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, M.D. & Ph.D., Principal Investigator — 1st Affiliated Hospital, Sun Yat-Sen University; Jianbo Liang, M.D., Principal Investigator — 2nd Affiliated Hospital, Guangzhou Medical College; Yunhua Liao, M.D., Principal Investigator — 1st Affiliated Hospital, Guangxi Medical University; Xinzhou Zhang, M.D. & Ph.D., Principal Investigator — Shenzhen People's Hospital; Fei Xiong, M.D., Principal Investigator — Wuhan No.1 Hospital; Hao Zhang, M.D., Principal Investigator — 3rd Xiangya Hospital, Central South University; Ping Fu, M.D. & Ph.D., Principal Investigator — West China Hospital; Yonggui Wu, M.D.& Ph.D., Principal Investigator — 1st Affiliated Hospital, Anhui Medical University; Minghui Zhao, M.D.&Ph.D., Principal Investigator — Peking University First Hospital; Xuewang Li, M.D., Principal Investigator — Peking Union Medical College Hospital; Li Hao, MD, Principal Investigator — 2nd Affiliated Hospital, Anhui Medical University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China